CLINICAL TRIAL: NCT02355301
Title: How to Improve the Quality of Care in Patients With Orthopaedic Disorders? - by Using the ICF in All Patients After Conservative or Surgical Treatment. - Through the Creation of an International Norm to Improve the Surgical Precision
Brief Title: Improve the Quality of Care in Patients With Orthopaedic Disorders
Acronym: QualOrtho
Status: Recruiting | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Orthopeadic team in Saint-luc Hospital Brussels (Unknown); Université Catholique de Louvain (Other); Institute of Mechanics, Materials and Civil Engineering UCL (Unknown)
Responsible Party: Principal Investigator, Detrembleur, Professor, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Other Study IDs: CD26012015
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Orthopedic Disorder
Keywords: ICF, impairment, activity, satisfaction, quality of care
MeSH Terms: conditions — Musculoskeletal Diseases; Motor Activity; Personal Satisfaction | interventions — Orthopedic Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with orthopedic disorders: Patients with muscular skeletal impairments receiving a treatment (A, B, C...). The investigators compare these treatments (A, B, C...) in function of ICF model in order to improve the quality of care in orthopedic department.
  Interventions: Procedure: orthopedic

INTERVENTIONS:
Procedure: orthopedic — Compare the type of treatment chosen by the orthopedist with a functional assessment (ICF-WHO model)

SUMMARY:
The main objective of the investigators is to improve the quality of care in patients with orthopedic disorders followed in St Luc hospital (Brussels Belgium). To do this, the investigators want to assess the impact of Orthopedic treatments at the structural level (bone structure, muscle, etc.), at the functional level (mobility, strength, stiffness...), on the restriction of activities of patients (walking, make its care daily..) and on the limitation of participation in the life of every day (sport, work, social life, cultural...). This functional evaluation of patients with orthopedic disorders by the ICF model is an original approach rarely used in muscular-skeletal impairments that can very improve the management of these patients and their quality of life. In addition, the investigators associate the harvesting of all medical and computer data collected by high-precision tools in the surgical treatments, to better define the surgical precision and improve the quality of surgical care.

DETAILED DESCRIPTION:
The investigators will recruit patients with orthopedic disorders on voluntary basis through department in St Luc Hospital in Brussels, old of 0 to 90 years, men and women with muscular-skeletal impairments (arthrosis, bone or muscle injury, ....). The investigators will exclude patients with multiple pathologies or not able to understand the instructions. They thus impropre the effectiveness of the treatment in Orthopaedics by better defining the route of most effective surgical first for the patient in arthroplasty (mini invasive, posterior, anterior), the most appropriate knee prosthesis type (design of prothesis), the conservative treatment properly to improve the quality of life of patients with orthopedic disorders (plaster, brace, physiotherapy...). They will evaluate the impact of treatments at the structural level (bone structure, muscle, etc.), at the functional level (mobility, strength, stiffness...), on the restriction of activities of patients (walking, make its care daily..) and on the limitation of participation in the life of every day (sport, work, social life, cultural...) following the ICF-WHO model.

In addition, they will dispose of data necessary to better define the surgical precision (international organization for standardization ISO Norm), the quality of surgical care by analyzing data collected by high-precision tools at the surgical treatments.

Patients will be subject to different clinical assessments, fill out questionnaires or come to the laboratory for analysis of the movement depending on the goal defined for each patient. Patients will have their current clinical follow-up (RX, scanner, mobility, force measurement, stiffness...) which the investigators be able to join a quantified analysis of the movement in the laboratory, satisfaction questionnaires, questionnaires measuring the impact of treatment on quality of life and their restriction of activities. It is a broad-spectrum study to try to improve the quality of care within a service target of orthopedics.

ELIGIBILITY:
Inclusion Criteria:

* all patients with orthopedic disorders : muscular skeletal impairment

Exclusion Criteria:

Dementia patients with multiple disorders Patients who do not understand the instructions

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with orthopedic disorders usually followed in the Department of Orthopedics clinics (St Luc Hospital - Brussels - Belgium)
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-04-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
activities | 6 months
  improve the gait; improve the daily activities (washing, eating, dressing...)

SECONDARY OUTCOMES:
Impairment: ICF domain | 6 months
  force, stiffness, mobility, dexterity
participation: ICF domain | 6 months
  effect of treatment on Sports, work, cultural and associative life

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Cornu, MD,PhD, Principal Investigator — Cliniques universitaires St Luc Brussels
Locations (1):
- Cliniques universitaires St Luc Brussels, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Caty GD, Detrembleur C, Bleyenheuft C, Deltombe T, Lejeune TM. Effect of upper limb botulinum toxin injections on impairment, activity, participation, and quality of life among stroke patients. Stroke. 2009 Jul;40(7):2589-91. doi: 10.1161/STROKEAHA.108.544346. Epub 2009 Apr 30. PMID 19407231
- [Result] Bollens B, Gustin T, Stoquart G, Detrembleur C, Lejeune T, Deltombe T. A randomized controlled trial of selective neurotomy versus botulinum toxin for spastic equinovarus foot after stroke. Neurorehabil Neural Repair. 2013 Oct;27(8):695-703. doi: 10.1177/1545968313491002. Epub 2013 Jun 10. PMID 23757297